CLINICAL TRIAL: NCT06421428
Title: Urinary Incontinence: Lived Experience of Adult Women. A Phenomenological Study
Brief Title: Living With Urinary Incontinence: Women's Experiences in a Qualitative Phenomenological Study
Acronym: LEI
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Sara Trapani, Principal Investigator, Midwife (RM), PhD student, IRCCS San Raffaele
Other Study IDs: LEI
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence; Experience, Life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women's single sample: The population under investigation will be made up of women aged ≥ 18 years (excluding pregnant women and women who have given birth less than 40 days) suffering from urinary incontinence and who understand and speak in the Italian language. Will be enrolled on a voluntary basis women who have already had at least a couple of pelvic floor rehabilitation meetings at the outpatient clinic of the San Raffaele Hospital in Milan, within the time frame foreseen by the study, because they are also able to narrate their experience of re-education of the pelvic floor.
  Interventions: Other: LEI Interview; Other: LEI Survey

INTERVENTIONS:
Other: LEI Interview — In accordance with the IPA (Interpretative phenomenological analysis) methodology, a semi-structured interview outline will be defined, aimed at understanding the lived experiences of women ("lived experience") during their coexistence with urinary incontinence and during the treatment process.
  The screwdriver questions were formulated starting from the scientific literature and with reference to the Theoretical Domains Framework (TDF), created and validated by Michie et al. (2005) and later updated by Cane et al. (2012). The interview questions will be discussed in a focus group composed of a uro-gynecologist, two midwives, a nurse, an expert in qualitative methodology. The final screwdriver questions resulting from the focus group will be tested on a small group of women.
Other: LEI Survey — Some sociodemographic data identified from the reference literature will be collected in paper form immediately at the end of each interview, for the description of the sample. The data will concern: age, nationality, marital status, level of education, number of children, menopause, social relationships, level of information, period of onset of symptoms, type of symptomatology, frequency of episodes of urinary incontinence, quantity of urinary leakage, uro-gynecological pathological history.

SUMMARY:
Study Description: Scientific literature demonstrated the negative influence of Urinary Incontinence (UI) on the quality of life connected to the physical, psychological, and social health of women.

However, a limited number of studies investigated in depth the emotional experience of women affected by this disorder, their behaviors, and their experiences in managing the problem. Health professionals need to understand these aspects to offer the best care, also taking into account women's cultural and territorial differences. Research conducted on the topic in the Italian context is lacking, therefore the present study aims to explore, in a Northern Italian context, the experience of adult women affected by UI.

Study Design: Qualitative phenomenological study (observational, cross-sectional, monocenter) Objective: To explore, in a Northern Italian context, the experience of women aged ≥ 18 years affected by Urinary Incontinence (UI) Study Population: Women ≥ 18 years old, not pregnant nor having given birth for less than 40 days, suffering from urinary incontinence who access the Pelvic Floor Rehabilitation Outpatient Clinic of the San Raffaele Hospital in Milan.

Sample Size: Women who have already had at least a couple of pelvic floor rehabilitation meetings at the outpatient clinic of the San Raffaele Hospital in Milan, within the time frame foreseen by the study. These subjects represent a precious resource and are considered "more informative for the researcher" as they testify to the emotions and daily life that influence the symptoms of urinary incontinence, but they are also able to narrate their experience of re-education of the pelvic floor.

It is assumed that approximately 20 women will be involved to reach data saturation.

Statistical Design: The interviews will be analyzed with the hermeneutic-phenomenological IPA (Interpretative phenomenological analysis) method, which involves the identification of units of meaning, categories and themes in accordance with the language of the speakers. The analysis of qualitative data will be made possible thanks to the use of data management software (NViVO). The socio-demographic data collected will be presented with absolute and relative frequencies

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age ≥ 18 years old
3. Urinary Incontinence
4. Informed consent signed
5. Comprehension of written and spoken Italian language
6. Female patients of the pelvic floor rehabilitation outclinic at San Raffaele Hospital

Exclusion Criteria:

1. Male sex
2. Young age (< 18 years)
3. Pregnancy
4. Puerperium (up to 40 days post-partum)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population under investigation will be made up of women aged ≥ 18 years (excluding pregnant women and women who have given birth less than 40 days) suffering from urinary incontinence and who understand and speak in the Italian language. Will be enrolled on a voluntary basis women who have already had at least a couple of pelvic floor rehabilitation meetings at the outpatient clinic of the San Raffaele Hospital in Milan, within the time frame foreseen by the study, because they are also able to narrate their experience of re-education of the pelvic floor.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
LEI (Lived Experience Incontinence) Interview | Baseline
  To explore, in a Northern Italian context, the experience of women aged ≥ 18 years affected by Urinary Incontinence (UI) through a semi-structured interview (open questions).
  Specifically, the topics addressed in the interview will be:
  * Emotions and daily life of women with UI (i.e. subjective meaning of UI, lifestyle changes, women's mood)
  * Behavioral strategies implemented to deal with the problem (i.e. choice to give up leisure activities, society's attention to the problem, tools and sources of information)
  * Perceptions regarding UI treatment plan (i.e. health expectations and desires, decision-making process that led to undertaking the treatment)

SECONDARY OUTCOMES:
LEI (Lived Experience Incontinence) survey | Baseline
  To collect some sociodemographic data regarding women affected by UI: age, nationality, marital status, level of education, number of children, menopause, social relationships, level of information, period of onset of symptoms, type of symptomatology, frequency of episodes of urinary incontinence, quantity of urinary leakage, uro-gynecological pathological history.

CONTACTS AND LOCATIONS:
Overall Officials: Duilio F. Manara, Study Chair — Director of Center for Nursing Research and Innovation (CeNRI); Massimo Candiani, Study Chair — Director of U.O. Obstetrics and Gynecology; Stefano Salvatore, Study Chair — U.O. Obstetrics and Gynecology; Stefania Rinaldi, Study Chair — U.O. Obstetrics and Gynecology; Ilaria Baini, Study Chair — U.O. Obstetrics and Gynecology; Giulia Villa, Study Chair — Center for Nursing Research and Innovation (CeNRI); Sara Trapani, Principal Investigator — U.O. Obstetrics and Gynecology
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No